CLINICAL TRIAL: NCT00664352
Title: A Double Blind, Placebo Controlled Trial to Investigate the Efficacy and Safety of Two Concentrations of Juvidex (Mannose-6-Phosphate) in Accelerating the Healing of Split Thickness Skin Graft Donor Sites Using Different Dosing Regimes
Brief Title: Juvidex (Mannose-6-Phosphate) in Accelerating the Healing of Split Thickness Skin Graft Donor Sites
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Dr Jim Bush, Renovo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1004-0082
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Wound
Keywords: Double blind; Placebo controlled; wound healing
MeSH Terms: conditions — Wounds and Injuries | interventions — mannose-6-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Mannose-6-Phosphate (Juvidex)
- 2 (Experimental)
  Interventions: Drug: Mannose-6-Phosphate (Juvidex)
- 3 (Experimental)
  Interventions: Drug: Mannose-6-Phosphate (Juvidex)
- 4 (Experimental)
  Interventions: Drug: Mannose-6-Phophate (Juvidex)
- 5 (Other)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mannose-6-Phosphate (Juvidex) — * 100µL of 300mM (8.46 mg/100μL) Juvidex will be injected intradermally into each cm2 of one 3cm2 donor site and into the 0.5cm border around the donor site no more than 20 minutes before graft harvest (total dose 750µL). A further 300µL of 300mM (8.46 mg/100μL) Juvidex will be applied topically within 30 minutes of graft harvest and 24 hours after graft harvest.
  * 100µL of placebo will be injected intradermally into each cm2 of the other 3cm2 donor site and into the 0.5cm border around the donor site no more than 20 minutes before graft harvest (total dose 750µL). A further 300µL of placebo will be applied topically within 30 minutes of graft harvest and 24 hours after graft harvest.
  Arms: 1
Drug: Mannose-6-Phosphate (Juvidex) — * 100µL of 600mM(16.93 mg/100μL) Juvidex will be injected intradermally into each cm2 of one 3cm2 donor site and into the 0.5cm border around the donor site no more than 20 minutes before graft harvest (total dose 750µL). A further 300µL of 600mM (16.93 mg/100μL) Juvidex will be applied topically within 30 minutes of graft harvest and 24 hours after graft harvest.
  * 100µL of placebo will be injected intradermally into each cm2 of the other 3cm2 donor site and into the 0.5cm border around the donor site no more than 20 minutes before graft harvest (total dose 750µL). A further 300µL of placebo will be applied topically within 30 minutes of graft harvest and 24 hours after graft harvest.
  Arms: 2
Drug: Mannose-6-Phosphate (Juvidex) — * 300µL of 300mM (8.46 mg/100μL) Juvidex will be applied topically to one 3cm2 donor site within 30 minutes of graft harvest and 24 hours after graft harvest.
  * 300µL of placebo will be applied topically to the other 3cm2 donor site within 30 minutes of graft harvest and 24 hours after graft harvest.
  Arms: 3
Drug: Mannose-6-Phophate (Juvidex) — * 300µL of 600mM (16.93 mg/100μL) Juvidex will be applied topically to one 3cm2 donor site within 30 minutes of graft harvest and 24 hours after graft harvest.
  * 300µL of placebo will be applied topically to the other 3cm2 donor site within 30 minutes of graft harvest and 24 hours after graft harvest.
  Arms: 4
Drug: Placebo — * 100µL of placebo will be injected intradermally into each cm2 of one 3cm2 donor site and into the 0.5cm border around the donor site no more than 20 minutes before graft harvest (total dose 750µL). A further 300µL of placebo will be applied topically within 30 minutes of graft harvest and 24 hours after graft harvest.
  * Standard Care (moist wound healing dressings alone) will be applied to the other 3cm2 donor site.
  Arms: 5

SUMMARY:
The objective of this study is to compare the efficacy of two concentrations of Juvidex with placebo on the healing of split thickness skin graft donor sites

DETAILED DESCRIPTION:
Split thickness skin grafting is the transplantation of a patient's own cutaneous tissue harvested from an area of normal skin, to replace an area of skin loss or injury. The split thickness skin graft (SSG) is one of the most commonly performed operations in plastic and reconstructive surgery1. Indications for split skin grafting include: reconstruction after the surgical removal of cutaneous malignancies, to replace tissue lost in full-thickness burns and to cover chronic non-healing cutaneous ulcers. As with all grafting procedures, a donor site wound is created, and, in the case of SSGs, the wound is a partial-thickness wound that heals by re-epithelialisation. Often, the graft donor site is the slowest to heal, and it is the source of most of the postoperative discomfort. In patients who have sustained major burns affecting large percentages of their cutaneous surface area, early closure of burn wounds with autologous skin grafts can be limited by the lack of adequate donor sites. These donor sites may need to be re-harvested to provide further skin cover; however a delay of 2 to 3 weeks is often required to allow these sites to heal prior to re-harvesting.

A treatment to accelerate the healing of SSG donor sites produced after harvest would address an area of high medical need, not only by providing an area available for re-harvest, but also by reducing the potential associated morbidities to the patient including pain and infection. This could also reduce length of hospital stay with associated reduced healthcare costs.

Transforming growth factor betas (TGF-beta), are a naturally occurring protein which plays a central role in the wound healing response. Juvidex is being developed by Renovo as a therapeutic agent administered to accelerate the healing of acute wounds. The proposed mechanism of action is antagonistic and involves inhibiting the activation of TGF-beta 1 and TGF beta 2.

Using healthy volunteers is an ideal way of studying the healing process on split thickness skin graft donor sites since the donor sites can be created so that they are exactly anatomically matched. These matched pairs can then be used to compare drug against placebo.

The trial is being undertaken to assess the effects of intradermally injected and topically applied Juvidex on the healing of small skin graft donor sites in volunteer subjects. The trial will also compare the effects of a placebo treatment with standard care alone in the healing of the donor sites. This will enable any placebo effect to be accurately measured and allow an accurate assessment of actual drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-85 years who have given written informed consent.
* A body mass index between 18-35 calculated using Quetelets index-weight (kg)/height² (m).
* Subjects with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests and ECG as specified in the trial protocol (see Protocol Section 6.4.2). All laboratory tests must be performed within 28 days of the first trial dose administration.
* Female patients of child bearing potential who are using a highly effective method(s) of contraception and agree to do so from at least the screening visit until one month after administration of the final study dose. For the purposes of the protocol, highly effective method(s) of contraception will be defined as consistently and correctly used implants, injectables, combined oral contraceptives, sexual abstinence or a vasectomised partner

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have history or evidence of hypertrophic or keloid scarring.
* Subjects with tattoos, birthmarks, moles or previous scars within 3cm of the area to be investigated during the trial.
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring.
* Subjects who have had surgery in the area to be investigated within one year of the first dosing day.
* Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Subjects with any clinically significant medical condition or history of any condition that would impair wound healing including :

  * Subjects with renal impairment (creatinine clearance (CLcr) of 80/ml/min or less)
  * Significant hepatic impairment (LFTs >3 times upper limit of normal).
  * Congestive heart failure with a classification of >2 according to the NYHA Classification (see appendix 5).
  * A history of myocardial infarction, ischaemic heart disease (or presenting with symptoms or signs compatible with ischaemic heart disease), coronary vasospasm or peripheral vascular disease.
  * Subjects, with significant cerebrovascular disease including a history of stroke, transient ischaemic attacks or haemorrhage.
  * Malignancy (unless treated and disease-free for 5 years).
  * Autoimmune disease (including active rheumatoid arthritis), immunosuppression (oral corticosteroids) or chemotherapy within the last 12 months.
  * Uncontrolled hypertension SBP > 180 mmHg, DBP > 95mmHg.
  * Diabetes (except diet controlled)
  * Significant respiratory disease.
* Subjects with a history of clinically relevant allergy, hypersensitivity, angioedema, or anaphylaxis.
* Subjects with a progressive neurological condition including Parkinson's disease, Alzheimer's disease and uncontrolled epilepsy.
* Subjects with a known history of chronic viral infection (Hepatitis, HIV) or ongoing active infection.
* Subjects with bleeding disorders including haemophilia, purpura or thrombocytopenia or receiving anticoagulants (e.g. warfarin, coumadin).
* Subjects who have taken any investigational product in the twelve months prior to first trial dose administration.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects with a history of substance abuse or dependency ( a history of recreational use of cannabis is acceptable assuming a negative urine test for cannabis at screen. Subjects who have had a history of alcohol abuse but have been dependency free for 12 months will still be eligible).
* Subjects with any condition or serious illness which, in the opinion of the Investigator, would interfere with participation in the study.
* Subjects with an ongoing psychiatric condition requiring treatment or psychosis (including depression with psychosis, bipolar disease and schizophrenia).
* Female subjects who are breast feeding, or intending to become pregnant or breast feed during the study period (subjects must be using adequate contraception and have a negative pregnancy test at screening - see Inclusion).
* Female subjects who have had any change in their oral contraceptive medication (if applicable) in the 2 months prior to screening, or anticipate any change during study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The time to complete wound closure as assessed by the investigating physician | Measured up to Day 28

SECONDARY OUTCOMES:
Local wound tolerability | Up to Day 28 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB. MRCS, Principal Investigator — General Medical Council
Locations (1):
- 09Clinical Trials Unit, Renovo Limited, Manchester, United Kingdom